CLINICAL TRIAL: NCT00449046
Title: Clinical Assessment of GW815SF Salmeterol/Fluticasone Propionate (HFA MDI) in Pediatric Patients With Bronchial Asthma -A Long Term (24-week) Study-
Brief Title: Clinical Assessment Of GW815SF Salmeterol/Fluticasone Propionate(HFA MDI) In Pediatric Patients With Bronchial Asthma -A Long Term (24-week) Study-
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110101
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Bronchial Asthma
Keywords: salmeterol/fluticasone propionate combination; pediatric bronchial asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: GW815SF Salmeterol/Fluticasone propionate(HFA MDI)

SUMMARY:
This study evaluates the long-term (24-week) safety and efficacy of GW815SF Salmeterol/fluticasone propionate(HFA MDI) 50/100mcg(administered as 2 inhalations of 25/50mcg) bid in pediatric patients with bronchial asthma.

ELIGIBILITY:
Inclusion criteria:

* Inclusion Criteria for Entry in Run-in Period

A pediatric patient already diagnosed as having bronchial asthma who meets all of the following criteria is eligible for the study:

* Male or female patients aged ≥5 and ≤14 years. Enrolment of a female patient of childbearing potential is allowed only if she is tested negative in the pregnancy testing at the start of treatment period and if she agrees to undergo pregnancy testing at the protocol-specified timings and to take contraceptive measures without fail during the study period.
* Written informed consent must be obtained from the legally acceptable representative of the subject. Consent of the subject him/herself should also be obtained, wherever possible, after giving an explanation in an as easy to understand as possible manner.
* An outpatient who has been treated with ICS (FP 100-200μg/day or equivalent) for at least 4 weeks prior to Visit 1.
* Is suitable, in the investigator's/subinvestigator's judgment, for treatment with GW815SF HFA MDI 25/50μg (administered as 2 inhalations of 25/50μg) bid.
* Able to use a peak flow meter in a correct manner in the investigator's/subinvestigator's judgment.
* Able to use MDI in a correct manner (with the assistance of his/her caregiver as necessary) in the investigator's/subinvestigator's judgment.

Inclusion Criteria for Entry in Treatment Period A subject will be considered eligible for inclusion in the treatment period only if he/she has completed the run-in period and meets the following criterion.

1. Has been able, in the investigator's/subinvestigator's judgment, to make entries in the asthma diary and measure PEF, as directed, during the run-in period.

Exclusion criteria:

* Exclusion Criteria for Entry in Run-in Period

A patient who applies any of the following criteria is not eligible for the study:

* Admitted to the hospital due to asthma exacerbation within 8 weeks prior to Visit 1.
* Used systemic steroid within 4 weeks prior to Visit 1.
* Received antibacterials or antivirals for treatment of upper or lower respiratory tract infection within 2 weeks prior to Visit 1.
* Has a safety problem in participation in the study because of a serious, uncontrolled systemic disease including nervous system disorder.
* Has or is suspected to have deep-seated mycosis or infection to which no effective antibacterial agent is available.
* Has or is suspected to have hypersensitivity to the investigational product, rescue medication or any ingredients of them.
* Is pregnant or lactating, may be pregnant, or plans for pregnancy during the study period.
* Has received the last dose in another clinical study within 2 months prior to this study.
* Is not eligible for the study in the investigator's/subinvestigator's judgment.

Exclusion Criteria for Entry in Treatment Period

A subject who applies to any of the following criteria is not eligible for the study:

1. Admitted to the hospital due to asthma exacerbation during the run-in period.
2. Had upper or lower respiratory tract infection during the 2 weeks just before Visit 2.
3. Used prohibited drugs during the 2 weeks just before Visit 2.
4. Is not eligible for the study in the investigator's/subinvestigator's judgment.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (3):
- Japan (3):
  - GSK Clinical Trials Call Center, Funabashi, Chiba
  - GSK Clinical Trials Call Center, Setagaya, Tokyo
  - GSK Clinical Trials Call Center, Takasaki, Gunma

RESULTS

PARTICIPANT FLOW:
Groups:
- Salmeterol/Fluticasone Propionate: Salmeterol/fluticasone propionate patients received 2 inhalations twice daily each inhalation was 25/50mcg for 24 weeks(Total daily dose was 100/200mcg)
Period: Overall Study
Arm/Group | Salmeterol/Fluticasone Propionate
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (2.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants] — One participant counted twice due to having multiple races.
  participants
    Asian | 39
    White | 1

OUTCOME MEASURES:

1. Primary Outcome: Most Frequent Adverse Events - On Therapy
Description: Adverse events, Clinical laboratory tests, Adrenocortical function test, Physical examinations, 12-lead electrocardiogram (ECG), Oropharyngeal examination were included.
Time Frame: Baseline to Week 24
Population: Safety analysis was performed on the primary outcome measures, adverse events and on the safety population defined as all subjects who entered the treatment period and received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Participants
  Laryngopharyngitis | 8
  Bronchitis | 8
  Nasopharyngitis | 8
  Asthma | 8
  Pharyngitis | 6
  Pyrexia | 5
  Otitis media | 4
  Pharyngotonsillitis | 3
  Laryngotracheo bronchitis | 3
  Molluscum contagiosum | 3
  Stomatitis | 3

2. Primary Outcome: Serious Adverse Events (SAEs) - On Therapy
Description: Number of participants considered by the investigator to be related to study medication.
  Adverse events, Clinical laboratory tests, Adrenocortical function test, Physical examinations, 12-lead ECG, Oropharyngeal examination were included. Frequency threshold of reported SAE's is 0%(100% reported)
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Participants | 1

3. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF) During Weeks 1-24
Description: PEF taken daily and average used for week 1-24 value. The peak expiratory flow rate measures how fast a person can (exhale) air. Then, compares it to normal flow rates to predict obstruction and disease. The average PEF for a child or adolescent whose height is 43" is 147 L/min, whose height is 66" is 454 L/min.
Time Frame: Baseline and during Weeks 1-24
Population: Efficacy analyses were performed on the secondary outcome measures and Full analysis set, defined as all the subjects who entered the treatment period, excluding all those who received no dose of study medication or who had no post-baseline data.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
L/min | 32.9 (34.48)

4. Secondary Outcome: Change From Baseline in Percent Predicted Morning Peak Expiratory Flow (PEF) During Weeks 1-24
Description: Percent Predicted Morning Peak Expiratory flow were the percent of patients that were predicted to have their Peak expiratory flow in the morning.
Time Frame: Baseline and during Weeks 1-24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Percent Change | 12.50 (11.294)

5. Secondary Outcome: Change From Baseline in Evening Peak Expiratory Flow (PEF) During Weeks 1-24
Description: The peak expiratory flow rate measures how fast a person can (exhale) air. Then compares it to normal flow rates to predict obstruction and disease. The average PEF for a child or adolescent whose height is 43" is 147 L/min, whose height is 66" is 454 L/min.
Time Frame: Baseline and during Weeks 1-24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
L/min | 31.2 (29.28)

6. Secondary Outcome: Change From Baseline in Circadian Variation in Peak Expiratory Flow (PEF) During Weeks 1-24
Description: Circadian Variation means the various changes in a day. The peak expiratory flow rate measures how fast a person can (exhale) air using a mini-Wright peak flow meter. The average PEF for a child or adolescent whose height is 43" is 147 L/min, whose height is 66" is 454 L/min.
Time Frame: Baseline and during Weeks 1-24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Percent Change | -1.62 (3.583)

7. Secondary Outcome: Number of Participants With Symptom-Free Nights and Days
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Participants
  Baseline | 29
  Week 24 | 31

8. Secondary Outcome: Number of Participants With Rescue Medication-Free Nights and Days
Description: Rescue free means without the use of other medication.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 40
Participants
  Baseline | 33
  Week 24 | 32

ADVERSE EVENTS:
Arm/Group | Salmeterol/Fluticasone Propionate
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 40
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Salmeterol/Fluticasone Propionate
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Salmeterol/Fluticasone Propionate
Laryngopharyngitis (Infections and infestations) | 8/40
Bronchitis (Infections and infestations) | 8/40
Nasopharyngitis (Infections and infestations) | 8/40
Asthma (Respiratory, thoracic and mediastinal disorders) | 8/40
Pharyngitis (Infections and infestations) | 6/40
Pyrexia (General disorders) | 5/40
Otitis Media (Infections and infestations) | 4/40
Pharyngotonsillitis (Infections and infestations) | 3/40
Laryngotracheo bronchitis (Infections and infestations) | 3/40
Molluscum contagiosum (Infections and infestations) | 3/40
Stomatitis (Gastrointestinal disorders) | 3/40
Gastroenteritis (Infections and infestations) | 2/40
Sinusitus (Infections and infestations) | 2/40
tonsillitus (Infections and infestations) | 2/40
Acetonaemic vomiting (Gastrointestinal disorders) | 2/40
Abdominal pain (Gastrointestinal disorders) | 2/40
Heat Rash (Skin and subcutaneous tissue disorders) | 2/40
Eczema (Skin and subcutaneous tissue disorders) | 2/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.